CLINICAL TRIAL: NCT00912600
Title: A Prospective Multicenter Study Examining the Criteria That Determine ICU Admission of Patients Over 80 Who Present to an Emergency Department and Evaluating the Impact of ICU Admission on Short and Mid-term Vital and Functional Outcome
Brief Title: Intensive Care Unit (ICU) Admission Decisions in the Elderly : the ICE-CUB Study
Acronym: IceCub
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Other Study IDs: AOR 03 035
Record Dates: First submitted 2009-06-02; First posted 2009-06-03 (Estimated); Last update posted 2012-07-26 (Estimated); Status verified 2009-05

CONDITIONS: Patient Admission; Death; Activities of Daily Living
Keywords: Intensive Care Units; Triage; Aged, 80 and over; Death; Activities of Daily Living; Health Services Research; Health Care Quality, Access, and Evaluation
MeSH Terms: conditions — Death

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: Elderly individuals presenting to one of 15 emergency departments and possibly qualifying for admission to an ICU
  Interventions: Other: Intensive Care Unit admission

INTERVENTIONS:
Other: Intensive Care Unit admission — Intensive Care Unit admission

SUMMARY:
Percentage of patients over 80 admitted in ICU varies greatly from one center to another. ICU admission criteria of older patients are scarcely described and benefit of ICU admission for those patients is uncertain. In this study, we prospectively studied old patients arriving to the emergency department of 15 French hospitals with conditions that potentially warrant ICU admission.The working hypothesis was that ICU admission was associated with a 20% decrease in six-month mortality.

DETAILED DESCRIPTION:
This was a prospective multicenter observational cohort study of elderly individuals presenting to one of 15 emergency departments and possibly qualifying for admission to an ICU. To be included, subjects had to be aged at least 80 years and be diagnosed by the ED physician with one of 74 conditions potentially warranting ICU admission.Outcome studied are ICU eligibility as assessed by emergency and ICU physicians, hospital and six-month death and changes in functional status in the six month following emergency department visit.

ELIGIBILITY:
Inclusion Criteria:

* Age over 80
* Be assigned by the emergency physician with one of 74 conditions potentially warranting ICU admission

Exclusion Criteria:

* Patient's refusal

Min Age: 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Old patients arriving to the emergency department of 15 French hospitals with conditions that potentially warrant ICU admission.
Sampling Method: Non-Probability Sample
Enrollment: 2643 (Actual)
Dates: Start 2004-11; Primary Completion 2006-01 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
ICU eligibility as assessed by emergency and ICU physicians | At the admission

SECONDARY OUTCOMES:
Hospital death | During the hospitalisation
Change in functional status | During 6 months
Six-month death | During 6 months after the end of the hospitalisation

CONTACTS AND LOCATIONS:
Overall Officials: Bertrand GUIDET, MD, Principal Investigator — Assistance Publique Hopitaux de Paris
Locations (1):
- Hôpital Saint-Antoine, Paris, France

REFERENCES:
- [Derived] Boumendil A, Angus DC, Guitonneau AL, Menn AM, Ginsburg C, Takun K, Davido A, Masmoudi R, Doumenc B, Pateron D, Garrouste-Orgeas M, Somme D, Simon T, Aegerter P, Guidet B; ICE-CUB study group. Variability of intensive care admission decisions for the very elderly. PLoS One. 2012;7(4):e34387. doi: 10.1371/journal.pone.0034387. Epub 2012 Apr 11. PMID 22509296